CLINICAL TRIAL: NCT02764294
Title: Effectiveness of the Distraction Methods on Pain, Anxiety and Satisfaction During Cystoscopy
Brief Title: Effectiveness of the Distraction Methods During Cystoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Principal Investigator, Elif Gezginci, RN, PhD, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 50687469-1491-263-16/1648-736
Record Dates: First submitted 2016-05-04; First posted 2016-05-06 (Estimated); Last update posted 2019-03-07 (Actual); Status verified 2017-12

CONDITIONS: Pain; Anxiety; Satisfaction
Keywords: anxiety; pain; satisfaction; cystoscopy; music; video; stress ball; nursing
MeSH Terms: conditions — Pain; Anxiety Disorders; Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Music Group (Active Comparator): Music group was listened to a music of their choise with a headset. The music intervention was started about 10-15 minutes before cystoscopy and continued during the whole procedure. Types of music were Turkish folk music, Turkish art music, Turkish arabesque music, Turkish pop music, foreign pop music, rock music, and classical music.
  Interventions: Other: Music Group
- Stress Ball Group (Active Comparator): Stress ball group was given stress ball into both their palms about 10-15 minutes before cystoscopy. Participants were instructed to "squeeze the balls twice after counting up to five" and "repeat it until the end of the procedure".
  Interventions: Other: Stress Ball Group
- DVD Group (Active Comparator): DVD group was watched a DVD of their choice (documentaries, interesting and amazing videos, comedies) on a ceiling-mounted monitor positioned at a comfortable distance to the participant.
  Interventions: Other: DVD Group
- Control Group (No Intervention): Participants received usual care from health professionals. They didn't receive any intervention.

INTERVENTIONS:
Other: Music Group — Music group was listened to a music of their choise with a headset. The music intervention was started about 10-15 minutes before cystoscopy and continued during the whole procedure. Types of music were Turkish folk music, Turkish art music, Turkish arabesque music, Turkish pop music, foreign pop music, rock music, and classical music.
  Arms: Music Group
Other: Stress Ball Group — Music group was given stress ball into both their palms about 10-15 minutes before cystoscopy. Participants were instructed to "squeeze the balls twice after counting up to five" and "repeat it until the end of the procedure".
  Arms: Stress Ball Group
Other: DVD Group — DVD group was started to be watched a DVD of their choise about 10-15 minutes before cystoscopy and continued during the whole procedure.
  Arms: DVD Group

SUMMARY:
Cystoscopy is a pain procedure and patients may experience anxiety and dissatisfaction before and during the procedure. Especially male patients feel more pain than females during cystoscopy. The aim of this study is to compare effectiveness of three different distraction methods on pain, anxiety and satisfaction of the male patients during cystoscopy.

DETAILED DESCRIPTION:
Cystoscopy is a reliable and effective method used commonly to investigate tumors and pathological or suspicious views related to bladder and urethra. The patients may feel pain, anxiety and dissatisfaction when cystoscope is inserted into the bladder. Thus nonpharmacological and pharmacological methods are used to decrease pain, anxiety and dissatisfaction levels of the patients during the procedure. Music is the most commonly used distraction method during cystoscopy, but there are few studies in this issue (only music) on literature. In additon, there isn't any study related to stress ball use during cystoscopy and there isn't any study which comparatives effectiveness of the multiple distraction methods to reduce pain, anxiety and dissatisfaction levels during this procedure. Therefore the investigators aimed to compare effectiveness of three different distraction methods (music, stress ball and DVD) on pain, anxiety and satisfaction of the patients during cystoscopy.

ELIGIBILITY:
Inclusion Criteria:

* to be male and over 18 years old
* to be first csytoscopy
* to be rigid csytoscopy

Exclusion Criteria:

* to have a contradiction for csystoscopy (lidocaine allergies, urinary tract infection, no anatomical problems with the urethra etc.)
* to be used any analgesic drug at least 24 hours prior to cystoscopy
* to be made manipulations such as double j stent placement or removal, and bladder biopsy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Pain Measure | "5-10 minutes before", "during" and "5 minutes after" cytoscopy
  The average score change on pain intensity as measured by VAS scale.

SECONDARY OUTCOMES:
Anxiety Measure | "5-10 minutes before" and "5 minutes after" cytoscopy
  The average score change on anxiety level as measured by STAI-State Anxiety scale.
Satisfaction Measure | "5 minutes after" cytoscopy
  The average score change on satisfaction level as measured by STAI-State Anxiety scale.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Gezginci, RN, PhD, Principal Investigator — University of Health Sciences, Gulhane Training and Research Hospital, Department of Urology, Ankara, Turkey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aaronson DS, Walsh TJ, Smith JF, Davies BJ, Hsieh MH, Konety BR. Meta-analysis: does lidocaine gel before flexible cystoscopy provide pain relief? BJU Int. 2009 Aug;104(4):506-9; discussion 509-10. doi: 10.1111/j.1464-410X.2009.08417.x. Epub 2009 Feb 23. PMID 19239453
- [Background] Burke DM, Shackley DC, O'Reilly PH. The community-based morbidity of flexible cystoscopy. BJU Int. 2002 Mar;89(4):347-9. doi: 10.1046/j.1464-4096.2001.01899.x. PMID 11872022
- [Background] Cano-Garcia Mdel C, Casares-Perez R, Arrabal-Martin M, Merino-Salas S, Arrabal-Polo MA. Use of Lidocaine 2% Gel Does Not Reduce Pain during Flexible Cystoscopy and Is Not Cost-Effective. Urol J. 2015 Nov 14;12(5):2362-5. PMID 26571322
- [Background] Chen YT, Hsiao PJ, Wong WY, Wang CC, Yang SS, Hsieh CH. Randomized double-blind comparison of lidocaine gel and plain lubricating gel in relieving pain during flexible cystoscopy. J Endourol. 2005 Mar;19(2):163-6. doi: 10.1089/end.2005.19.163. PMID 15798411
- [Background] Ellerkmann RM, Dunn JS, McBride AW, Kummer LG, Melick CF, Bent AE, Blomquist JL. A comparison of anticipated pain before and pain rating after the procedure in patients who undergo cystourethroscopy. Am J Obstet Gynecol. 2003 Jul;189(1):66-9. doi: 10.1067/mob.2003.377. PMID 12861140
- [Background] Greenstein A, Greenstein I, Senderovich S, Mabjeesh NJ. Is diagnostic cystoscopy painful? Analysis of 1,320 consecutive procedures. Int Braz J Urol. 2014 Jul-Aug;40(4):533-8. doi: 10.1590/S1677-5538.IBJU.2014.04.13. PMID 25251958
- [Background] Gunendran T, Briggs RH, Wemyss-Holden GD, Neilson D. Does increasing hydrostatic pressure ("bag squeeze") during flexible cystoscopy improve patient comfort: a randomized, controlled study. Urology. 2008 Aug;72(2):255-8; discussion 258-9. doi: 10.1016/j.urology.2008.02.072. Epub 2008 Jun 12. PMID 18554699
- [Background] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Background] Hudson BF, Ogden J, Whiteley MS. Randomized controlled trial to compare the effect of simple distraction interventions on pain and anxiety experienced during conscious surgery. Eur J Pain. 2015 Nov;19(10):1447-55. doi: 10.1002/ejp.675. Epub 2015 Jan 30. PMID 25641687
- [Background] Kesari D, Kovisman V, Cytron S, Benjamin J. Effects on pain and anxiety of patients viewing their cystoscopy in addition to a detailed explanation: a controlled study. BJU Int. 2003 Nov;92(7):751-2. doi: 10.1046/j.1464-410x.2003.04477.x. PMID 14616460
- [Background] Kim JH, Park SY, Kim MG, Choi H, Song D, Cho SW, Song YS. Pain and satisfaction during rigid cystoscopic ureteral stent removal: a preliminary study. BMC Urol. 2014 Nov 18;14:90. doi: 10.1186/1471-2490-14-90. PMID 25406892
- [Background] Krajewski W, Koscielska-Kasprzak K, Rymaszewska J, Zdrojowy R. How different cystoscopy methods influence patient sexual satisfaction, anxiety, and depression levels: a randomized prospective trial. Qual Life Res. 2017 Mar;26(3):625-634. doi: 10.1007/s11136-016-1493-1. Epub 2017 Jan 3. PMID 28050795
- [Background] Li H, Cheng Y, Li J, Chen Y, Yuan J, Yang S, Shi H, Li W, Yang S, Wang W, Xu G, Zhao S. NaHCO3-Buffered Lidocaine Gel for Outpatient Rigid Cystoscopy in Men. J Perianesth Nurs. 2016 Apr;31(2):154-7. doi: 10.1016/j.jopan.2014.05.014. Epub 2016 Jan 8. PMID 27037169
- [Background] Raheem OA, Mirheydar HS, Lee HJ, Patel ND, Godebu E, Sakamoto K. Does Listening to Music During Office-Based Flexible Cystoscopy Decrease Anxiety in Patients: A Prospective Randomized Trial. J Endourol. 2015 Jul;29(7):791-6. doi: 10.1089/end.2015.0029. Epub 2015 Apr 13. PMID 25630866
- [Background] Soomro KQ, Nasir AR, Ather MH. Impact of patient's self-viewing of flexible cystoscopy on pain using a visual analog scale in a randomized controlled trial. Urology. 2011 Jan;77(1):21-3. doi: 10.1016/j.urology.2010.08.012. Epub 2010 Oct 25. PMID 20974485
- [Background] Stewart M, Cox-Davenport RA. Comparative Analysis of Registered Nurses' and Nursing Students' Attitudes and Use of Nonpharmacologic Methods of Pain Management. Pain Manag Nurs. 2015 Aug;16(4):499-502. doi: 10.1016/j.pmn.2014.09.010. Epub 2014 Dec 12. PMID 25499026
- [Background] Taghizadeh AK, El Madani A, Gard PR, Li CY, Thomas PJ, Denyer SP. When does it hurt? Pain during flexible cystoscopy in men. Urol Int. 2006;76(4):301-3. doi: 10.1159/000092051. PMID 16679829
- [Background] Wang DS. Re: Does Listening to Music during Office-Based Flexible Cystoscopy Decrease Anxiety in Patients: A Prospective Randomized Trial. J Urol. 2016 Feb;195(2):448-9. doi: 10.1016/j.juro.2015.10.153. Epub 2015 Nov 2. No abstract available. PMID 26853024
- [Background] Yerlikaya G, Laml T, Elenskaia K, Hanzal E, Kolbl H, Umek W. Pain perception during outpatient cystoscopy: a prospective controlled study. Eur J Obstet Gynecol Reprod Biol. 2014 Feb;173:101-5. doi: 10.1016/j.ejogrb.2013.11.007. Epub 2013 Nov 14. PMID 24300559
- [Background] Yeo JK, Cho DY, Oh MM, Park SS, Park MG. Listening to music during cystoscopy decreases anxiety, pain, and dissatisfaction in patients: a pilot randomized controlled trial. J Endourol. 2013 Apr;27(4):459-62. doi: 10.1089/end.2012.0222. Epub 2012 Dec 5. PMID 23009573
- [Background] Zhang ZS, Wang XL, Xu CL, Zhang C, Cao Z, Xu WD, Wei RC, Sun YH. Music reduces panic: an initial study of listening to preferred music improves male patient discomfort and anxiety during flexible cystoscopy. J Endourol. 2014 Jun;28(6):739-44. doi: 10.1089/end.2013.0705. Epub 2014 Mar 31. PMID 24548148